CLINICAL TRIAL: NCT04232254
Title: Defining Beef and Meal Frequency as Key Components of a Healthy Eating Pattern for Muscle Health and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: National Cattlemen's Beef Association, a contractor to the Beef Checkoff (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 20243
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-10

CONDITIONS: Meal Frequency; Dietary Habits; Muscle Protein Synthesis
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Animal Protein - Skewed Distribution (Active Comparator): Animal-based protein foods with 3 meals per day consisting of 10-, 30-, and 60% of dietary protein for breakfast, lunch, and dinner, respectively.
  Interventions: Behavioral: Animal-based Protein Foods; Behavioral: Skewed Protein Distribution
- Plant Protein - Skewed Distribution (Experimental): Plant-based protein foods with 3 meals per day consisting of 10-, 30-, and 60% of dietary protein for breakfast, lunch, and dinner, respectively.
  Interventions: Behavioral: Skewed Protein Distribution; Behavioral: Plant-based Protein Foods
- Animal Protein - Balanced Distribution (Experimental): Animal-based protein foods with 5 meals per day consisting of 20% of dietary protein per meal.
  Interventions: Behavioral: Animal-based Protein Foods; Behavioral: Balanced Protein Distribution
- Plant Protein - Balanced Distribution (Experimental): Plant-based protein foods with 5 meals per day consisting of 20% of dietary protein per meal.
  Interventions: Behavioral: Plant-based Protein Foods; Behavioral: Balanced Protein Distribution

INTERVENTIONS:
Behavioral: Animal-based Protein Foods — Participants will consume animal-based protein foods.
  Arms: Animal Protein - Balanced Distribution; Animal Protein - Skewed Distribution
Behavioral: Skewed Protein Distribution — Participants will consume 3 meals per day consisting of 10-, 30-, 60% of dietary protein for breakfast, lunch, and dinner, respectively.
  Arms: Animal Protein - Skewed Distribution; Plant Protein - Skewed Distribution
Behavioral: Plant-based Protein Foods — Participants will consume plant-based protein foods.
  Arms: Plant Protein - Balanced Distribution; Plant Protein - Skewed Distribution
Behavioral: Balanced Protein Distribution — Participants will consume 5 meals per day consisting of 20% of dietary protein per meal.
  Arms: Animal Protein - Balanced Distribution; Plant Protein - Balanced Distribution

SUMMARY:
Adopting a healthy eating pattern is important for meeting dietary recommendations and weight management. Although less clear, it seems reasonable to assume that the eating patterns we typically follow can also affect our psychological wellbeing. As such, healthy eating patterns are often adapted to suit one's personal preference. For example, many people choose to follow a vegetarian-style eating pattern whereby meat, poultry, and seafood are excluded from the diet. However, current research suggests that vegetarian eating patterns may result in decreased synthesis of new muscle proteins when compared to the typical meat-based US-style diet. This ultimately leads to reduced muscle quality and mass which increases the risk of dependence and mobility limitations later in life.

Another important factor to consider when adapting a healthy eating pattern is the frequency and distribution of meals throughout the day. In the US, protein intake is typically skewed throughout the day such that people consume more protein at dinner when compared to breakfast. This skewed distribution combined with a low meal frequency (3 meals per day) can also sacrifice the rate of muscle protein synthesis. As such, it is important to investigate the interaction between food choices, meal frequency, and protein distribution to promote muscle health and prevent development of disease and disability. In addition, it is also important to understand how these eating patterns affect enjoyment and pleasure following meals. This work will help to determine healthy eating patterns that promote muscle health and psychological wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-40
* Pre-menopausal
* Recreationally active
* Weight stable for prior 6 months
* Consumption of meat-based diet for >6 months

Exclusion Criteria:

* Age outside of range (20 - 40)
* Pregnancy
* Irregular menstrual cycles
* Participation in previous research using 2H2O or [13C6]phenylalanine
* Participation in other ongoing research that interferes with this study (e.g., conflicting diet, activity interventions, etc.)
* Any hospitalization or surgery for a metabolic, cardiovascular, or neuromusculoskeletal complication within the past year
* Allergy or hypersensitivity to local anesthetics, latex, or adhesives (bandages, medical tape, etc.)
* Excess scarring after injury
* History of excess bleeding after cut
* Chronic or frequent dizziness/fainting, and arm or leg weakness/numbness
* Arthritis
* Tumors
* Mental Illness
* Hepatorenal, cardiovascular musculoskeletal, autoimmune, or neurological disease or disorder
* Predisposition to hypertrophic scarring or keloid formation
* Physical activity limitations
* Consumption of ergogenic-levels of dietary supplements that may affect muscle mass (e.g., creatine, HMB), insulin-like substances, or anabolic/catabolic pro-hormones (e.g., DHEA) within 6 weeks prior to participation
* Consumption of thyroid, androgenic, or other medications known to affect endocrine function
* Consumption of medications known to affect protein metabolism (e.g., prescription-strength corticosteroids, nonsteroidal anti-inflammatories, or acne medication)
* Unwillingness to comply with study procedures
* Weight unstable (variation >5% of bodyweight in last 6-12 months)
* Pregnancy
* Allergy to dairy product or lactose intolerance
* Current or previous tobacco use with last 6 months
* Obesity (body mass index; BMI > 30 kg m-2)
* Score of less than 14 or greater than 24 on Godin-Shephard Leisure-Time Physical Activity Questionnaire

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Compare fractional synthesis rate of myofibrillar proteins to different dietary protein food sources and meal frequencies | Day 1 - Day 9
  Rate of building new protein in skeletal muscle contractile protein

SECONDARY OUTCOMES:
Valence (Pleasantness or Unpleasantness) | Immediately prior to workout, immediately post workout, and immediately post meal on habituation days 2, 4, and 6 and intervention days 3, 5, and 7
  Measurement of feelings of un/pleasantness via survey responses to a measure of valence (Feeling Scale)
Arousal (Alertness) | Immediately prior to workout, immediately post workout, and immediately post meal on habituation days 2, 4, and 6 and intervention days 3, 5, and 7
  Measurement of feelings of alertness to via survey responses to a measure of arousal (Felt Arousal Scale)
Arousal (Alertness) | Immediately prior to workout, immediately post workout, and immediately post meal on habituation days 2, 4, and 6 and intervention days 3, 5, and 7
  Measurement of feelings of alertness to via survey responses to a measure of arousal (Activation-Deactivation Adjective Check List).

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas A Burd, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers

REFERENCES:
- [Derived] Askow AT, Barnes TM, Zupancic Z, Deutz MT, Paulussen KJM, McKenna CF, Salvador AF, Ulanov AV, Paluska SA, Willard JW, Petruzzello SJ, Burd NA. Impact of Vegan Diets on Resistance Exercise-Mediated Myofibrillar Protein Synthesis in Healthy Young Males and Females: A Randomized Controlled Trial. Med Sci Sports Exerc. 2025 Sep 1;57(9):1923-1934. doi: 10.1249/MSS.0000000000003725. Epub 2025 Apr 4. PMID 40197715